CLINICAL TRIAL: NCT05822817
Title: A Prospective, Randomized Controlled Study to Compare the Effect of Sevoflurane and Propofol for Maintenance of Anesthesia on Postoperative Recovery After Transsphenoidal Resection of Pituitary Adenoma
Brief Title: Comparison of Postoperative Recovery of Sevoflurane and Propofol After Transsphenoidal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K3501
Record Dates: First submitted 2023-03-13; First posted 2023-04-21 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-04

CONDITIONS: Pituitary Adenoma
Keywords: Anesthesia; Transsphenoidal surgery; Enhanced recovery after surgery
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane (Experimental): Anesthesia is maintained with sevoflurane.
  Interventions: Drug: sevoflurane
- propofol (Experimental): Anesthesia is maintained with continuous infusion of propofol.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: sevoflurane — Anesthesia is maintained with inhalation of sevoflurane. The concentration of sevoflurane was adjusted to maintain anesthetic depth, aiming for a bispectral index of 40-60.
  Arms: sevoflurane
Drug: propofol — Anesthesia is maintained with an effect-site target-controlled infusion of propofol (2-6ug/ml) based on the Marsh mode. The concentration of propofol was adjusted to maintain anesthetic depth, aiming for a bispectral index of 40-60.
  Arms: propofol

SUMMARY:
Currently, total intravenous anesthesia (TIVA) and inhaled anesthesia are both commonly used for transsphenoidal pituitary adenoma resection. However, optimal choice for anesthesia maintenance in transsphenoidal surgery remains unclear. Previous studies focusing on this question provided fragmentary assessment and controversial results. The goal of this clinical trial is to investigate whether propofol and sevoflurane have different effect on post-anesthetic recovery after transsphenoidal resection of pituitary adenoma.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, aged from 18 to 70
2. American Society of Anesthesiologists (ASA) class I - III
3. Patients scheduled for transsphenoidal surgery requiring general anesthesia managed with endotracheal intubation

Exclusion Criteria:

1. Patients allergic or contraindicated to sevoflurane, propofol, or other drugs used during surgery
2. Severe pulmonary disease, saturation of peripheral oxygen (SpO2) < 90%
3. Severe nervous system disease with consciousness disorder
4. Patients scheduled for intensive care unit (ICU) after surgery
5. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
15-item quality of recovery score (QoR-15) | 24 hours after end of surgery
  The QoR-15 score ranges from 0 to 150 (higher is better). The investigators record the scores of two groups 1 day after the surgery.

SECONDARY OUTCOMES:
Time to awake from anesthesia | From stopping sevoflurane or propofol to awake, approximately 30 minutes
  The time between discontinuing drugs and response to verbal command.
Time to extubation | From stopping sevoflurane or propofol to recovery of spontaneous breathing and withdrawal of tracheal tube, approximately 30 minutes
  The time between discontinuing drugs and withdrawal of tracheal tube.
Agitation or sedation level during emergence | From stopping sevoflurane or propofol to complete awakening, approximately 30 minutes
  The highest Richmond agitation and sedation scale score (RASS) during emergence. The RASS score ranges from -5 to +4, and a lower score indicates a more sedative level.
Coughing and bucking during emergence | From stopping sevoflurane or propofol to complete awakening, approximately 30 minutes
  Coughing score ranges from 0 to 3, and a higher score indicates a severer outcome.The investigators record the highest coughing score during emergence.
Time to discharge from postanesthesia care unit (PACU) | From admit into PACU to discharge from PACU, approximately 45 minutes
  The time between admission into PACU and discharging from PACU with Aldrete score over 9. Aldrete score ranges from 0 to 10, and a higher score indicates a better recovery from anesthesia.
PACU antiemetic drug use | From admit into PACU to discharge from PACU, approximately 45 minutes
  The drug use due to postoperative nausea and vomiting in PACU.
PACU analgesic drug use | From admit into PACU to discharge from PACU, approximately 45 minutes
  The drug use due to postoperative pain in PACU.
Post operative nausea and vomiting score | 24 hours after end of surgery
  Score: 0, no nausea and vomiting; 1-4, mild nausea and vomiting; 5-6, moderate nausea and vomiting; 7-10, severe nausea and vomiting.
Concentration of serum adrenocorticotropic hormone (ACTH) | 24 hours after end of surgery
  The investigators examine the serum level of ACTH in pg/mL.
Concentration of serum cortisol | 24 hours after end of surgery
  The investigators examine the serum level of cortisol in ug/dL.
Concentration of serum thyroid-stimulating hormone (TSH) | 24 hours after end of surgery
  The investigators examine the serum level of TSH in uIU/mL.
Concentration of serum growth hormone (GH) | 24 hours after end of surgery
  The investigators examine the serum level of GH in ng/mL.
Concentration of serum gonadotrophin | 24 hours after end of surgery
  The investigators examine the serum level of gonadotrophin in IU/L.
Concentration of serum prolactin (PRL) | 24 hours after end of surgery
  The investigators examine the serum level of PRL ng/mL.
Counts of peripheral blood lymphocyte | 24 hours after end of surgery
Incidence of hypotension during anesthesia | From start of surgery to end of surgery, on an average of 2 hours
  Hypotension is defined as decrease of mean arterial pressure (MAP) more than 20% of baseline.
Incidence of hypertension during anesthesia | From start of surgery to end of surgery, on an average of 2 hours
  Hypertension is defined as increase of MAP more than 20% of baseline.
Time to discharge from hospital | From end of surgery to discharge from hospital, on an average of 2 days
  The time between end of surgery and discharge from hospital.

OTHER OUTCOMES:
Number of participants with postoperative complications | After the surgery till discharge
  The investigators record major postoperative complications and other complications related to anesthesia not mentioned above.
Number of participants with postoperative complications | After discharge till 7 days after the surgery
  The investigators record major postoperative complications and other complications related to surgery and anesthesia by telephone follow-up.
Numerical rating scale (NRS) pain score at postoperative day 7 | 7 days after the surgery
  The investigators record NRS pain score (0 to 10, higher the more painful) of patients on the 7th day after the surgery by telephone follow-up.
Post operative nausea and vomiting score at postoperative day 7 | 7 days after the surgery
  Score: 0, no nausea and vomiting; 1-4, mild nausea and vomiting; 5-6, moderate nausea and vomiting; 7-10, severe nausea and vomiting.
Sleep quality score at postoperative day 7 | 7 days after the surgery
  The investigators record the sleep quality score (0 to 10, higher the better) of patients on the 7th day after the surgery by telephone follow-up.
Appetite score at postoperative day 7 | 7 days after the surgery
  The investigators record the appetite score (0 to 10, higher the better) of patients on the 7th day after the surgery by telephone follow-up.
30-day readmission | At the 1st postoperative month
  The investigators record the patients' readmission to our hospital due to any pathological reason (to outpatient or inpatient).
Concentration of serum cortisol | At the 3rd postoperative month
  The investigators examine the serum level of cortisol in ug/dL.
Concentration of serum growth hormone (GH) | At the 3rd postoperative month
  The investigators examine the serum level of GH in ng/mL.
Concentration of serum gonadotrophin | At the 3rd postoperative month
  The investigators examine the serum level of gonadotrophin in IU/L.
Concentration of serum thyroid-stimulating hormone (TSH) | At the 3rd postoperative month
  The investigators examine the serum level of TSH in uIU/mL.
Concentration of serum prolactin (PRL) | At the 3rd postoperative month
  The investigators examine the serum level of PRL ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD, Study Chair — Department of Anesthesiology, Peking Union Medical College Hospital; Lulu Ma, MD, Study Director — Department of Anesthesiology, Peking Union Medical College Hospital; Bing Xing, MD, Principal Investigator — Department of Neurosurgery, Peking Union Medical College Hospital; Wei Lian, MD, Principal Investigator — Department of Neurosurgery, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cafiero T, Cavallo LM, Frangiosa A, Burrelli R, Gargiulo G, Cappabianca P, de Divitiis E. Clinical comparison of remifentanil-sevoflurane vs. remifentanil-propofol for endoscopic endonasal transphenoidal surgery. Eur J Anaesthesiol. 2007 May;24(5):441-6. doi: 10.1017/S0265021506002080. Epub 2007 Mar 12. PMID 17376252
- [Background] Ali Z, Prabhakar H, Bithal PK, Dash HH. Bispectral index-guided administration of anesthesia for transsphenoidal resection of pituitary tumors: a comparison of 3 anesthetic techniques. J Neurosurg Anesthesiol. 2009 Jan;21(1):10-5. doi: 10.1097/ANA.0b013e3181855732. PMID 19098618
- [Background] Kim DH, Min KT, Kim EH, Choi YS, Choi SH. Comparison of the effects of inhalational and total intravenous anesthesia on quality of recovery in patients undergoing endoscopic transsphenoidal pituitary surgery: a randomized controlled trial. Int J Med Sci. 2022 Jun 13;19(6):1056-1064. doi: 10.7150/ijms.72758. eCollection 2022. PMID 35813289
- [Derived] Feng Y, Zhang Y, Lian W, Xue Y, Ma M, Yu X, Guo X, Ma L, Xing B, Huang Y. A randomized controlled trial to compare the effects of sevoflurane and propofol for maintenance of anesthesia on postoperative recovery quality in patients undergoing transsphenoidal resection of pituitary adenoma. BMC Anesthesiol. 2025 Aug 4;25(1):392. doi: 10.1186/s12871-025-03263-z. PMID 40760415